CLINICAL TRIAL: NCT02551523
Title: A Prospective, Randomised, Controlled, Open-label, Non-inferiority Trial to Compare the Efficacy of Standard of Care Combination Antiretroviral Therapy With a Simplified Dolutegravir Monotherapy in Patients With a Primary HIV-1 Infection Under Suppressive Early Standard of Care Antiretroviral Therapy
Brief Title: Early Simplified: A Trial to Compare the Efficacy of Standard of Care Combination Antiretroviral Therapy With a Simplified Dolutegravir Monotherapy in Patients With a Primary HIV-1 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2015-0288
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Monotherapy; Dolutegravir; Primary HIV Infection; Treatment Efficacy
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dolutegravir monotherapy (Experimental): 92 patients will be simplified to once daily dolutegravir monotherapy.
  Interventions: Drug: Dolutegravir
- Standard of care combination antiretroviral therapy (Active Comparator): 46 patients will go on with standard of care combination antiretroviral therapy consisting of either a protease inhibitor or a non-nucleoside reverse transcriptase inhibitor or a integrase inhibitor in combination with two nucleoside reverse transcriptase inhibitors.
  Interventions: Drug: Standard of care combinational antiretroviral therapy

INTERVENTIONS:
Drug: Dolutegravir — 92 patients will be simplified to once daily dolutegravir monotherapy
  Arms: Dolutegravir monotherapy
Drug: Standard of care combinational antiretroviral therapy
  Arms: Standard of care combination antiretroviral therapy

SUMMARY:
Long term toxicity of combination antiretroviral therapy (cART) is a substantial contributor to morbidity and mortality in chronically infected HIV positive individuals. To date it is still debated, whether long term nucleoside reverse transcriptase inhibitors (NRTI's) -sparing regimens are practicable or even superior compared to standard of care cART in terms of efficacy, safety and tolerability. In addition, data about efficacy of integrase inhibitor (INSTI) based monotherapy is lacking. We aim at investigating the efficacy of standard of care combination antiretroviral therapy with a simplified dolutegravir monotherapy in patients with a primary HIV-1 infection under suppressive early standard of care antiretroviral therapy. Briefly, hundred-thirty-eight patients with a documented primary HIV1- infection (PHI) will be recruited from the Zurich Primary HIV-1 Infection Study (ZHPI), which is an open label, non-randomized, observational, single-center study (http://clinicaltrials.gov, ID 5 NCT00537966). All subjects formerly underwent early cART consisting of either a protease inhibitor (PI) or a non-nucleoside reverse transcriptase inhibitor (NNRTI) or a INSTI in combination with two NRTIs at the time point of enrolment in the ZPHI and must be under a fully suppressive ART (i.e., <50 copies/ml) for at least 48 weeks at the time point of randomisation. The primary end point is the proportion of individuals with a viral failure at week 48 or before.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature,
* All patients ≥18 years with a documented primary HIV-infection undergoing standard of care cART (i.e., one active drug from the class of either the PIs, or the NNRTIs, or the INSTIs, in combination with two active drugs from the class of NRTIs) with no previous structured treatment interruption and with a suppressed viral load (defined as 50 copies/ml) during the previous 48 weeks,
* Participant of the Swiss HIV Cohort Study

Exclusion Criteria:

* Patients not willing to sign the informed consent form,
* Presence of ≥1 major integrase inhibitor resistance associated mutation according to the Sanford algorithm1,
* History of ≥2 consecutive plasma viremia levels >400 copies/ml at least two weeks apart,
* Ongoing (i.e., replicating) hepatitis B virus infection,
* Hemoglobin < 10 g/dl (men) and < 9 g/dl (women) at the time of enrolment,
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception,
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-11; Primary Completion 2018-10 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals with a viral failure [defined as ≥2 plasma viremia levels >50copies/ml at least two weeks apart] at week 48 or before. | 48 weeks
  The study seeks primarily to determine the efficacy (i.e., proportion of patients with a viral failure [defined as ≥2 plasma viremia levels >50copies/ml at least two weeks apart] at week 48 or before) of a simplified monotherapy (i.e., DTG) compared to a standard of care HIV triple-therapy in patients with a PHI treated with early ART under long term suppressive ART for at least 48 weeks.

SECONDARY OUTCOMES:
Quantification of latent HIV-1 reservoir by measurement of proviral DNA and cell-associated RNA at baseline (time point of randomization), and at week 48 | Week48
Proportion of individuals with a CSF HIV-1 RNA <50copies/ml in the CSF at week 48 after treatment simplification. | Week 48
Proportion of patients with an adverse event at week 48. | Week 48
Proportion of patients with a severe adverse event at week 48. | Week 48
Time to viral failure (defined as ≥2 plasma viremia levels >50copies/ml at least two weeks apart) at week 48. | Week 48
Proportion of individuals with blips (defined as one viral load >50 and <400 copies/ml with a next viral load <50 copies/ml) at week 48. | Week 48
Change from baseline CD4+ cell count from baseline at week 48. | Week 48
Proportion of individuals with new onset of proximal tubular renal dysfunction at week 48. | Week 48
Creatinine clearance change from baseline at week 48. | Week 48
Lipidic profile changes from baseline at week 48. | Week 48
Proportion of individuals developing a new CDC-event at week 48. | Week 48
Proportion of individuals withdrawing consent at week 48. | Week 48
Proportion of individuals being lost to follow-up at week 48. | Week 48
Proportion of individuals switching assigned treatment for any cause at week 48. | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Dominique L Braun, MD, Principal Investigator — Division of Infectious Diseases and Hospital Epidemiology, University Hospital Zurich, University of Zurich
Locations (1):
- University Hospital Zurich, University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Braun DL, Turk T, Tschumi F, Grube C, Hampel B, Depmeier C, Schreiber PW, Brugger SD, Greiner M, Steffens D, De Torrente-Bayard C, Courlet P, Neumann K, Kuster H, Flepp M, Bertisch B, Decosterd L, Boni J, Metzner KJ, Kouyos RD, Gunthard HF. Noninferiority of Simplified Dolutegravir Monotherapy Compared to Continued Combination Antiretroviral Therapy That Was Initiated During Primary Human Immunodeficiency Virus Infection: A Randomized, Controlled, Multisite, Open-label, Noninferiority Trial. Clin Infect Dis. 2019 Oct 15;69(9):1489-1497. doi: 10.1093/cid/ciy1131. PMID 30601950